CLINICAL TRIAL: NCT06239805
Title: "Effectiveness of Molecular Quantum Resonance (QMR) in the Rehabiltative Treatment of Gonarthrosis"
Brief Title: Quantum Molecular Resonance (QMR) Rehabiltative Treatment of Knee Osteoarthritis
Acronym: QMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Collaborators: Teresa Paolucci (Unknown); Mirko Pesce (Unknown); Roberto Buda (Unknown); Andrea Pantalone (Unknown)
Responsible Party: Principal Investigator, Antonia Patruno, Associate Professor, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ud'A Chieti-Pescara
Record Dates: First submitted 2023-01-20; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Knee Pain Chronic
Keywords: pain; physical therapy; QMR; gonarthrosis; synovial fluid; monocytes
MeSH Terms: conditions — Pain; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental intensive group (Experimental): Experimental: intensive treatment
  Interventions: Device: QMR
- Control extensive group (Active Comparator): extensive treatment
  Interventions: Device: QMR
- control sham group (Sham Comparator): sham group
  Interventions: Device: QMR

INTERVENTIONS:
Device: QMR — A: Treated group (active medical device): intensive protocol B: Treated Group (active medical device): extensive protocol C: Sham/Control group (medical device off)
  Patients will be treated as follows:
  A- Treated Group: three sessions a week, for a total of 6 sessions, with one session lasting of 30 minutes. The session involves the application of electrodes (adhesive plates), and Q- glove Touch (frequency/intensity)
  B- Treated Group: two sessions a week, for a total of 8 sessions, lasting a 20 minute session. The session involves the application of electrodes (adhesive plates), e Q-Touch glove (frequency/intensity)
  C- Control/Sham group: three sessions a week, for a total of 6 sessions, lasting a 30 minute session. The session involves the application of electrodes (adhesive plates), e Q-Touch glove with device off.

SUMMARY:
Gonarthrosis (osteoarthritis of the knee (OA) is a chronic-degenerative disease, characterized by progressive joint damage up to disability that affects about 40% of people over 65 years of age. Its typical pathological changes, articular cartilage degradation, synovial inflammation and subchondral bone thickening, are responsible for the pain and disability of patients. It is now known that "biophysical stimulation" techniques represent a non-invasive therapy used in orthopedic practice to enhance the reparative and anabolic activities of the tissues through an anti-inflammatory and chondro-protective effect.The aim of the study will be to evaluate the anti-inflammatory effects and the relative mechanisms of action of the therapeutic interventions of the QMR technology (Molecular Quantum Resonance) in the treatment of gonarthrosis through the use of in vivo and in vitro models. This technology, supplied by Telea Electronic Engineering s.r.l., exploits non-ionizing high-frequency waves in the range between 4 and 64 MHz at low intensity delivered through alternating electric fields. For the in vivo study, a double-blind randomized controlled clinical trial will be conducted. Both male and female subjects, aged between 40 and 80 years, with knee pain both in the acute and chronic phase of gonarthosis, diagnosed on standard radiography, will be enrolled. Patients will be randomized into 2 groups treated with an intensive or extensive protocol, and a third untreated control group. They will be evaluated at T0 (before treatment), at T1 (end of QMR treatment), and at T2 (one month after the end of treatment (follow-up)). All patients will be assessed for pain and functionality, furthermore synovial fluid and blood sampling will be performed, for the quantitative assessment of the inflammatory state considering the levels of the main pro-inflammatory cytokines and the pro/anti-inflammatory macrophage phenotype. In parallel, in order to delineate the molecular and cellular mechanism of action of QMR stimulation in vitro, a monocyte cell model (THP-1 cell line) will be used to evaluate the response of QMR treatment after treatment with known pro-inflammatory stimuli .

DETAILED DESCRIPTION:
For the in vivo study, a double-blind randomized controlled clinical trial will be conducted. Both male and female subjects, aged between 40 and 80 years, with knee pain both in the acute and chronic phase of gonarthosis, diagnosed on standard radiography, will be enrolled. Patients will be randomized into 2 groups treated with an intensive or extensive protocol, and a third untreated control group. They will be evaluated at T0 (before treatment), at T1 (end of QMR treatment), and at T2 (one month after the end of treatment (follow-up). All patients will be assessed for pain and functionality, furthermore synovial fluid and blood sampling will be performed, for the quantitative assessment of the inflammatory state considering the levels of the main pro-inflammatory cytokines and the pro/anti-inflammatory macrophage phenotype.

ELIGIBILITY:
Inclusion Criteria:

Both male and female subjects, aged between 40 and 80 years, with knee pain both in acute and chronic phase due to gonarthosis diagnosed on standard radiography will be enrolled.

* Diagnosis of gonarthrosis with VAS >3
* Presence of acute or chronic pain (the sample will be stratified in one phase next)
* Radiographic picture of gonarthrosis and staging score according to Kellegren-Lawrence classification (I-II-III)

Exclusion Criteria:

favism, hemolytic anemia

* severe hyperthyroidism - Graves' disease;
* drug treatment with Tapazole;
* thrombocytopenia less than 50,000 and serious coagulation disorders;
* severe cardiovascular instability;
* coagulation defects;
* alcohol abuse;
* hemochromatosis;
* patients being treated with food-nutraceutical supplements;
* pregnancy and bed rest;
* psychiatric pathologies;
* less than three months from previous knee infiltrations
* septic arthritis and/or febrile states
* anamnestic contraindications to the instrumental physical therapy in use (tumor pathologies past)

Furthermore, the following subjects will be excluded from the study:

* with rheumatic and autoimmune diseases
* patients with recent history of trauma and/or knee (ligament) sprain injuries

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Knee pain | T0 - 0 days
  Visual Analogue Scale (VAS)
Knee pain | T1 - 1 mounth of treatment
  Visual Analogue Scale (VAS)
Knee pain | T2 - 1 mounth after the end of treatment
  Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Function | T0 - 0 days
  Knee injury and Osteoarthritis Outcome Score (KOOS-I)
  - Lysholm Knee Scoring Scale
Function | T1 - 1 mounth of treatment
  Knee injury and Osteoarthritis Outcome Score (KOOS-I)
  - Lysholm Knee Scoring Scale
Function | T2 - 1 mounth after the end of treatment
  Knee injury and Osteoarthritis Outcome Score (KOOS-I)
  - Lysholm Knee Scoring Scale

OTHER OUTCOMES:
Kinesiophobia | T0 - 0 days
  Tampa Scale of Kinesiophobia - TSK
Kinesiophobia | T1 - 1 mounth of treatment
  Tampa Scale of Kinesiophobia - TSK
Kinesiophobia | T2 - 1 mounth after the end of treatment
  Tampa Scale of Kinesiophobia - TSK

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Patruno, PhD, Principal Investigator — University G. d'Annunzio Chieti Pescara
Locations (1):
- Don Orione Foundation, Pescara, PE, Italy

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.